CLINICAL TRIAL: NCT04200703
Title: Quality Improvement Center on Domestic Violence in Child Welfare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas (Other)
Collaborators: Futures Without Violence (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UKansas
Record Dates: First submitted 2019-09-25; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Multiple Forms of Child Abuse; Domestic Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Implementation of the Adult and Survivor Centered Approach.
  Interventions: Other: Adult and Child Survivor Centered Approach
- Comparison (No Intervention): No implementation of intervention.

INTERVENTIONS:
Other: Adult and Child Survivor Centered Approach — Child welfare workers and supervisors, and community partners will be trained in the Adult and Child Survivor Centered Approach, and supervisors will receive ongoing coaching and training.
  Arms: Intervention

SUMMARY:
The Quality Improvement Center on Domestic Violence in Child Welfare (QIC-DVCW) is a five-year federal cooperative agreement with the Children's Bureau to test an approach to improve how child welfare agencies and their partners work collaboratively to help families experiencing domestic violence. The safety and well-being of child survivors of domestic violence and child maltreatment are closely connected to the safety and well-being of the adult survivor of domestic violence. For this reason, the QIC-DVCW is testing an Adult & Child Survivor-Centered Approach to addressing the needs of both the parent and child, which includes effectively engaging and working with the person causing them harm. The following four research questions were developed to guide the work of the Recipient's evaluation of the QIC-DVCW, and Provider's data will help to answer these questions:

1. Does a collaborative, adult and child survivor-centered approach-that includes safely engaging and establishing accountability of the DV offender-improve adult and child survivor safety, child permanence, and child and family well-being for child welfare involved families experiencing DV?
2. For which families and in which social contexts does an adult and child survivor-centered approach improve these outcomes?
3. What factors are associated with successful implementation and sustainability of an adult and child survivor-centered approach?
4. What are the costs associated with the implementation and maintenance of an adult and child survivor-centered approach, and how do these costs compare to the costs of "practice as usual"?

ELIGIBILITY:
There are several aspects to study. Data collection strategies have distinct eligibility criteria. These are described below.

1. Overall Study

   Inclusion Criteria:

   Staff members of child welfare agencies and community partners, and the families experiencing domestic served in the intervention and comparison sites.

   Exclusion Criteria:

   All non-staff members of child welfare agencies and community partners, and the families experiencing domestic served in the intervention and comparison sites.
2. Caseworker, Supervisor, Community Partner Self-Survey

   Inclusion Criteria:

   Staff members of child welfare agencies and community partners in the intervention and comparison sites.

   Exclusion Criteria:

   All non-staff members of child welfare agencies and community partners in the intervention and comparison sites.
3. Caseworker Case Specific Survey

Inclusion Criteria:

Caseworkers (i.e., case carrying) in the intervention and comparison sites.

Exclusion Criteria:

Anyone who is not a caseworker in the intervention and comparison sites.

Inclusion Criteria by case. The following criteria must be met to be included in case-specific survey:

1. Newly investigated cases (i.e., cases that have been screened in for a response - investigation, alternate response - within the research period, in other words, not cases that have been open for DV for a while with no recent new reports)
2. Subject to investigation or alternative response
3. Active DV Cases (defined by type - partner violence and time -within the last year - of violence/cc
4. All survivors (inclusive of all gender identities)
5. Only if survivor whereabouts are known
6. Only families with at least one child that is or under 10 years old
7. Served by standard (i.e., not adolescent or youth units)
8. All relationships included (i.e., no type of relationship excluded)

4. Adult Survivor Survey

Inclusion criteria: Adult survivors of domestic violence who are part of a case that met the criteria of case specific survey and a case specific survey has been completed on that case.

Exclusion criteria: Anyone who is not an adult survivor of domestic violence and/or are not part of a case that met the criteria of case specific survey and/or a case specific survey has not been completed on that case.

5. People Who Use Violence web-based survey

Inclusion criteria: People who use violence who are part of a case that met the criteria of case specific survey and a case specific survey has been completed on that case.

Exclusion criteria: People who do not use violence and/or who are not part of a case that met the criteria of case specific survey and/or a case specific survey has not been completed on that case.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-29 (Estimated); Study Completion 2021-09-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline child safety at 6 months | Baseline and six months later
  Administrative data: maltreatment report, type of maltreatment
Change from baseline child residence permanency at 6 months | Baseline and six months later
  Administrative data: residence stability measured by type of residence and time in care
Change from baseline child education stability at 6 months | Baseline and six months later
  projected created items on surveys; caseworker survey and survey of parent (adult survivor) report of frequency of changes in educational setting, frequency of suspensions/expulsions
Change from baseline child exposure to domestic violence at 6 months | Baseline and six months later
  projected created items on surveys; caseworker survey and survey of parent (adult survivor); report of exposure
Change from baseline child social and emotional abilities at 6 months | Through study completion, an average of 1 year
  projected created items on surveys; caseworker survey and survey of parent report of perception of social and emotional abilities
Change from baseline child emotional and social development at 6 months | Through study completion, an average of 1 year
  projected created items on surveys; caseworker survey and survey of parent; report of perception of child's emotional and social development
Change from baseline child physical health at 6 months | Baseline and six months later
  projected created items on surveys; caseworker survey and survey of parent; report of perception of child's physical health
Change from baseline child supportive relationships with specific individuals at 6 months | Baseline and six months later
  projected created items on surveys; caseworker survey and survey of parent; report of child's supportive relationships
Change from baseline person who uses violence use of domestic violence/coercive control | One time point (retrospective pre and post) and Baseline and six months later
  projected created items on surveys; self-report of person using violence and adult survivor report of violence; frequency and type of violence used
Change of person who uses violence understanding of the nature, and dynamics, and impact of DV on adult and child survivors | One time point (retrospective pre and post) and Baseline and six months later
  projected created items on surveys; self-report of person using violence and adult survivor report
Change person who uses violence blaming adult survivor and justification for violence | One time point (retrospective pre and post) and Baseline and six months later
  projected created items on surveys; self-report of person using violence and adult survivor report
Change person who uses violence understanding of healthy relationships | One time point (retrospective pre and post) and Baseline and six months later
  projected created items on surveys; self-report of person using violence and adult survivor report
Change person who uses violence positive parent-child interactions | One time point (retrospective pre and post) and Baseline and six months later
  projected created items on surveys; self-report of person using violence and adult survivor report
Change from baseline adult survivor safer and more stable conditions at 6 months | Baseline and six months later
  projected created items on surveys; self-report adult survivor report of violence - frequency and type of violence used, assessment of risk level of violence, employment and housing stability
Change from baseline adult survivor social, cultural, and spiritual connections at 6 months | Baseline and six months later
  projected created items on survey, self-report by adult survivor
Change from baseline adult survivor resilience and growth mindset at 6 months | Through study completion, an average of 1 year
  projected created items on survey,, self-report by adult survivor
Change from baseline adult survivor nurturing parent-child interactions at 6 months | Baseline and six months later
  projected created items on survey, self-report by adult survivor
Change from baseline adult survivor social and emotional abilities at 6 months | Baseline and six months later
  projected created items on survey, self-report by adult survivor

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Carlson, PhD, Principal Investigator — University of Kansas School of Social Welfare
Locations (1):
- Juliana Carlson, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: No